CLINICAL TRIAL: NCT03460574
Title: How Can Change of Dysfunctional Expectations in Major Depression be Enhanced? An Experimental Study Targeting Cognitive Immunization
Brief Title: Targeting Cognitive Immunization in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-39k
Record Dates: First submitted 2018-01-29; First posted 2018-03-09 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Participants are assigned to one of four experimental groups in parallel for the duration of the study
Who Masked: Investigator
Masking Description: The investigator randomly assigns participants to one of the experimental conditions. Participants are not aware which experimental condition they are allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- INFORMATION (Experimental): Participants in this condition receive a manipulation suggesting that the performance test "TEMINT", they previously worked on, has been shown to be highly relevant for daily life and professional success. We anticipated that after receiving this fake information about the TEMINT, it would be difficult for participants to engage in cognitive immunization processes because the validity and utility of the expectation-disconfirming experience is explicitly highlighted.
  Interventions: Behavioral: INFORMATION
- SALIENCE (Experimental): Participants in this condition are asked to think about how well they performed on this really difficult performance test. We anticipated that this manipulation would enhance expectation change, as the salience of the expectation-disconfirming experience was explicitly increased.
  Interventions: Behavioral: SALIENCE
- ATTENTION (Experimental): Before working on the performance test, participants in this conditions receive the instruction to attentionally focus on their personal result in the performance test. Further, they are asked to specify what would be personally good result for them. We anticipated that after receiving this instruction, the expectation-disconfirming performance feedback should be salient for the participants, hence making it difficult for them to engage in cognitive immunization strategies.
  Interventions: Behavioral: ATTENTION
- CONTROL (Experimental): Participants in this condition receive no further information. Therefore, they are passing through the standard procedure of the previously developed experimental paradigm.
  Interventions: Behavioral: CONTROL

INTERVENTIONS:
Behavioral: INFORMATION — After receiving expectation-disconfirming positive performance feedback, participants receive standardized information that stresses the relevance of this experience. In particular, participants are told that the performance test they worked on is highly relevant for both professional success and personal life satisfaction.
  Arms: INFORMATION
Behavioral: SALIENCE — After receiving expectation-disconfirming positive performance feedback, partcipants in this condition are instructed to remember how well they performed on the performance test. Using a visual analogue scale, they were asked to specify how they performed relative to the other participants.
  Arms: SALIENCE
Behavioral: ATTENTION — Before working on the performance test, participants are instructed to pay attention to the feedback they receive. In particular, they are asked to enter what would be a personally good result for them. It is supposed that this shift of attention increases the salience of the expectation-disconfirming feedback.
  Arms: ATTENTION
Behavioral: CONTROL — This group does not receive any further intervention. Instead, participants of this group pass through the standard procedure of the EXPEC paradigm.
  Arms: CONTROL

SUMMARY:
Research has shown that people suffering from MDD tend to maintain dysfunctional expectations despite experiences that disconfirm expectations. Recently, it has been shown that this persistence of expectations is due to maladaptive information processing involving "cognitive immunization". This experimental study aims at testing three different strategies to inhibit cognitive immunization, in order to enhance expectation change.

DETAILED DESCRIPTION:
It appears adaptive to change one's expectations when continuously gaining expectation-disconfirming experiences; however, research has shown that people suffering from MDD have difficulty in changing their expectations after experiences that disconfirm expectations. Recently, the investigators have shown that this persistence of expectations is due to maladaptive information processing involving "cognitive immunization", defined as a cognitive reappraisal of expectation-disconfirming experiences in such a way that the individual's expectations are maintained. In view of psychotherapeutic interventions aiming to modify patients' dysfunctional expectations, effective strategies to inhibit cognitive immunization strategies need to be identified. Therefore, the aim of this study was to compare different immunization-inhibiting strategies with regard to their effectivity in enhancing expectation change. For this purpose, the investigators use a standardized experimental paradigm, which was developed and validated in a previous study.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of Major Depressive Disorder
* at least 18 years old
* sufficient German language knowledge

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Performance Expectations Scale - generalized | Directly prior to the performance test and directly after completing the performance test
  Change from Baseline to Postassessment in generalized performance expectations

SECONDARY OUTCOMES:
Performance Expectations Scale - task-specific | Directly prior to the performance test and directly after completing the performance test
  Change from Baseline to Postassessment in task-specific performance expectations

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kube, M. Sc., Principal Investigator — Philipps University Marburg
Locations (1):
- Schoen Klinik Bad Arolsen, Bad Arolsen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Background] Kube T, Rief W, Gollwitzer M, Glombiewski JA. Introducing an EXperimental Paradigm to investigate Expectation Change (EXPEC). J Behav Ther Exp Psychiatry. 2018 Jun;59:92-99. doi: 10.1016/j.jbtep.2017.12.002. Epub 2017 Dec 12. PMID 29253640